CLINICAL TRIAL: NCT02164617
Title: Development and Evaluation of an Evidence-based Intervention Guideline of the Wheelchair-bound Senior Elastic Band (WSEB) Exercise Program for the Demented Seniors in Long-term Care Facilities
Brief Title: Wheelchair-bound Senior Elastic Band (WSEB) Exercise Program for the Demented Seniors
Acronym: WSEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-2012-01-02(II); NSC-102-2314-B-037-054-MY2 (Other Grant/Funding Number: National Science Council)
Record Dates: First submitted 2014-06-10; First posted 2014-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Dementia
Keywords: Dementia; Wheelchair-bound seniors; Long-term care facilities; Elastic band exercise; Functional fitness; Daily life function; Depression; Problem behaviors
MeSH Terms: conditions — Dementia; Depression; Problem Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wheelchair-bound Senior Elastic Band (Experimental): Wheelchair-bound Senior Elastic Band (WSEB) exercise program has three phases: 1) warm-up: 6 movements to loosen up the body and elevate the energy for a safe transition to the next phase, 2) aerobic motions: 6 low-to-medium speed exercises to enhance the cardiovascular-respiratory workout, and 3) static stretching: 6 low-speed, gentle stretching exercises to build up muscle power/endurance and increase range of motion and flexibility. It is conducted three times per week, 40 minutes per practice.
  Interventions: Other: Wheelchair-bound Senior Elastic Band exercise program (WSEB)
- control (No Intervention): routine care

INTERVENTIONS:
Other: Wheelchair-bound Senior Elastic Band exercise program (WSEB) — Wheelchair-bound Senior Elastic Band exercise program (WSEB) three times per week, 40 minutes per practice
  Arms: Wheelchair-bound Senior Elastic Band

SUMMARY:
The goals of this three-year research project were: 1) to develop and evaluate the feasibility of the Wheelchair-bound Senior Elastic Band (WSEB) for the demented, wheelchair-bound seniors in long-term care facilities, 2) to evaluate the long-term effects of the instructor-led WSEB on the functional fitness, daily life function, depression, and problem behaviors of this senior population, and 3) to test the feasibility, compliance, and effectiveness of the DVD-led WSEB on this senior population.

DETAILED DESCRIPTION:
A three-year, longitudinal, triangulation research method was applied. First Year (Phase I): A preliminary WSEB, including hard copy descriptions and DVD demonstrations of each exercise, were sent to the 12 experts in the Delphi advisory panel for their critique and evaluation. First Year (Phase II): A quasi-experimental, one-group, pretest-posttest design was used to pilot-test the feasibility of the WSEB on a group of 15-20 demented, wheelchair-bound seniors in long-term care facilities. Second Year: A quasi-experimental, pre-post tests, non-equivalent control group design was used to test the long-term effects of the instructor-led WSEB on the functional fitness (cardiovascular-respiratory function, body flexibility, range of the joint's motion, and muscle strength and endurance), daily life function, depression, and problem behaviors of the demented, wheelchair-bound seniors in long-term care facilities. Eight long-term care facilities with 150 demented, wheelchair-bound seniors from southern Taiwan were recruited and randomly assigned based on the facilities to a WSEB experimental group or a waiting-list control group. Participants in the experimental group received the WSEB lead by the pre-trained and certified instructors, three times per week, 40 minutes per practice for 24 weeks; participants in the waiting-list control group remained regular activities in the facilities. One pre-test and two post-tests, 12 weeks apart, were conducted. Third Year: Using the same method as in the second year, participants from the second year were continued practicing the WSEB, but guided by a DVD, for another 36 weeks. The feasibility, compliance, and effectiveness of the DVD-led WSEB on the demented, wheelchair-bound seniors in long-term care facilities were tested, and another three post-tests, 12 weeks apart, were conducted on the same outcome measurements as in the second year.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 and over
* diagnosed with dementia by a physician or screened by the Mini-Mental State Examination (MMSE) as dementia
* wheelchair-bound seniors
* living in the long-term care facility for at least three months

Exclusion Criteria:

* having severe and acute cardiovascular, musculoskeletal, or pulmonary illnesses
* suffering from spinal cord injury with no rehabilitation potential

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functional fitness at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  1. Functional Fitness 1.1 Cardiovascular-Respiratory Function 1.1.1 Blood Pressure Digital Sphygmomanometer (OMRON - HEM707) 1.1.2 Lung Capacity TruZoneTM Peak Flow Meter 1.2 Body Flexibility 1.2.1 Upper Body Flexibility Back Scratch Test 1.2.2 Lower Body Flexibility Chair Sit-and-Reach Test 1.3 Range of the Joint's Motion 1.3.1 Flexion of the Shoulder Joint Goniometry 1.3.2 Abduction of the Shoulder Joint Goniometry 1.4 Muscle Strength and Endurance 1.4.1 Hand-Grip Strength Digital Handgrip Dynamometer (TKK - 5101) 1.4.2 Arm Muscle Endurance Arm Curl Test

SECONDARY OUTCOMES:
Change from baseline in daily life function at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  measured by Barthel Index (BI)
Change from baseline in depression at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  measured by Cornell Scale for Depression in Dementia Chinese version (CSDD)
Change from baseline in problem behaviors at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  Clifton Assessment Procedures for the Elderly-Behavior Rating Scale Chinese version (CAPE-BRS)

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Chen MC, Chen KM, Chang CL, Chang YH, Cheng YY, Huang HT. Elastic Band Exercises Improved Activities of Daily Living and Functional Fitness of Wheelchair-bound Older Adults with Cognitive Impairment: A Cluster Randomized Controlled Trial. Am J Phys Med Rehabil. 2016 Nov;95(11):789-799. doi: 10.1097/PHM.0000000000000518. PMID 27149585